CLINICAL TRIAL: NCT01138124
Title: Risk of Pancreatic Cancer and Renal Cancer in Patients Exposed to Gabapentin in the United Kingdom General Practice Research Database
Brief Title: Gabapentin and Risk of Pancreatic Cancer and Renal Cancer (GPRD)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114427; EPI40634 (Other: GSK); WEUSKOP4774 (Other: GSK)
Record Dates: First submitted 2010-06-03; First posted 2010-06-07 (Estimated); Results first posted 2011-01-07 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Renal Pelvis Cancer; Restless Legs Syndrome; Epilepsy; Neuropathic Pain; Chronic Pancreatitis; Hypertension; Pancreatic Cancer; Diabetes; Renal Cancer; Renal Cell Carcinoma
Keywords: renal cell carcinoma; epidemiology; pancreatic cancer; renal cancer; renal pelvis cancer; GPRD; case-control; Gapabentin
MeSH Terms: conditions — Restless Legs Syndrome; Epilepsy; Neuralgia; Pancreatitis, Chronic; Hypertension; Pancreatic Neoplasms; Diabetes Mellitus; Kidney Neoplasms; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- UK GPRD 1993-2008: The study cohort from which cases and controls are drawn is all subjects in the United Kingdom (UK) General Practice Research Database (GPRD) 1993-2008. Each member of the UK population is registered with a General Practice, which centralizes the medical information not only from the general practitioners themselves but also from specialist referrals and hospital attendances. Over 487 General Practices contribute data to the GPRD. Entry into the study cohort begins Jan 1, 1993 for all those who are registered in GPRD before that time, and at the time of registration if later than Jan 1, 1993.
  Interventions: Drug: Gabapentin prescriptions

INTERVENTIONS:
Drug: Gabapentin prescriptions — The exposure of interest is gabapentin use as defined by prescriptions recorded by the GPRD general practitioner (British National Formulary codes). Data on prescriptions for gabapentin will be extracted for each case and control from entry into the study cohort up to the index date (the exposure window). Gabapentin exposure will be parameterized as follows: (1) Ever versus never exposed; (2) Number of prescriptions; (3) Duration of exposure; and (4) Cumulative dose. These parameterizations will also be examined with a 2 year lag time from the index date, limiting the exposure window from entry into the study cohort up to 2 years prior to the index date.

SUMMARY:
High doses of gabapentin are associated with pancreatic acinar cell tumors in rats, but there has been no post marketing pancreatic carcinogenicity signal with gabapentin as reported by spontaneous reports in the Adverse Events Reporting System or in the published literature. In a published case-control screening study of the association of gabapentin with 55 cancers, the only cancer that met the screening criteria for possibly increased cancer risk with gabapentin exposure was renal (including renal pelvis) cancer. This association was judged to be likely due to or substantially accentuated by confounding by cigarette smoking, hypertension, and lifestyle (Cancer Causes Control 2009;20:1821-1835).

The primary objective of this study is to determine whether exposure to gabapentin is associated with an increased risk of developing pancreatic cancer or renal cancer in the United Kingdom (UK) General Practice Research Database (GPRD). Almost all members of the UK population are registered with a General Practice, which centralizes the medical information not only from the general practitioners themselves but also from specialist referrals and hospital attendances. Over 487 General Practices contribute data to the GPRD.

The study cohort from which cases and controls are drawn is all subjects in the GPRD 1993-2008. Gabapentin was approved in the UK in May 1993. Entry into the study cohort begins Jan 1, 1993 for all those who are registered in GPRD before that time, and at the time of registration if later than Jan 1, 1993. Patients with a first diagnosis of the respective cancer 1995-2008 are risk set matched with up to 10 controls within the same General Practice for age at cohort entry (within two years), sex, and year of entry into the study cohort (within one year). For cases, the index date is the date of first diagnosis of the respective cancer. The index date for controls is set as the date at which the follow-up time from cohort entry is the same as the case. The index date is chosen so as to give the control equal follow-up time to that of the case for ascertainment of use of gabapentin. Cases and controls will be required to have at least 2 years of follow-up in the study cohort before their index date. Data on gabapentin prescriptions are obtained for cases and controls from study cohort entry to the index date.

Crude and adjusted odds ratios and 95% confidence intervals (CI) will be produced from conditional logistic regression models, with additional analyses evaluating for latency and dose-response. For pancreatic cancer, covariates are smoking, body mass index, diabetes, epilepsy, neuropathic pain, and chronic pancreatitis. For renal cancer, covariates are smoking, body mass index, diabetes, hypertension, diuretic use, epilepsy, and neuropathic pain.

DETAILED DESCRIPTION:
Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymised and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice. Actual number of patients could be less than , as it is possible for a patient to be represented in more than one of the four arms (See "Participant Flow: Overall Study" Table) because of the risk set sampling.

ELIGIBILITY:
Inclusion Criteria:

* The study cohort from which cases and controls are drawn is all subjects in the UK GPRD 1993-2008. Entry into the study cohort begins Jan 1, 1993 for all those who are registered in GPRD before that time, and at the time of registration if later than Jan 1, 1993. Follow-up ends Dec 31, 2008, or earlier if the respective cancer is diagnosed, or if the subject leaves the GPRD for any reason including death.

Exclusion Criteria:

* Cases and controls will be required to have at least 2 years of follow-up in the study cohort before their index date (For cases, the index date is the date of first diagnosis of the respective cancer. The index date for controls is set as the date at which the follow-up time from cohort entry is the same as the case.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort from which cases and controls are drawn is all subjects in the UK GPRD 1993-2008. Entry into the study cohort begins Jan 1, 1993 for all those who are registered in GPRD before that time, and at the time of registration if later than Jan 1, 1993. Follow-up ends Dec 31, 2008, or earlier if the respective cancer is diagnosed, or if the subject leaves the GPRD for any reason including death. There are several advantages to the GPRD dataset for this study. It is a large dataset with detailed longitudinal prescription data, and long term follow-up (mean 7 years) to allow for latency in carcinogenicity. It provides good representation of the elderly who are disproportionately affected by pancreatic and renal cancers, and routinely includes data recorded by general practitioners on potential risk factors such as smoking and body mass index.
Sampling Method: Probability Sample
Enrollment: 54202 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were not recruited for nor enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and used to develop a patient cohort. All diagnoses and treatment are recorded in the course of routine medical practice.
Pre-assignment Details: Actual number of patients may be less, as it is possible for a patient to be represented in more than one of the four arms (See "Participant Flow: Overall Study" Table) because of the risk set sampling.
Groups:
- Pancreatic Cancer Cases: Incident pancreatic cancer, defined as first time pancreatic cancer diagnosis (READ/ Oxford Medical Information System [OXMIS] codes) in the General Practice Research Database (GPRD) study cohort. Entry into the GPRD study cohort began Jan 1, 1993, or at the time of GPRD registration if after Jan 1, 1993. Subjects were required to have at least 2 years of follow-up prior to the index date. The index date for cases was the date of incident pancreatic cancer diagnosis. Exocrine pancreatic cancer, endocrine pancreatic cancer, and carcinoma in situ were included. Cancer metastatic to the pancreas was excluded.
- Pancreatic Cancer Controls: Pancreatic cancer cases were risk set matched with up to 10 controls for sex, age at GPRD study cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site.
  The index date for controls was set as the date at which the follow-up time from cohort entry was the same as the case. The index date was chosen so as to give the control equal follow-up time to that of the case for ascertainment of use of gabapentin.
- Renal Cancer Cases: Incident renal cancer, defined as first time renal cancer diagnosis (READ/OXMIS codes) in the GPRD study cohort. Entry into the GPRD study cohort began Jan 1, 1993, or at the time of GPRD registration if after Jan 1, 1993. Subjects were required to have at least 2 years of follow-up prior to the index date. The index date for cases was the date of incident renal cancer diagnosis. Renal cell carcinoma and renal pelvis cancer were included; Wilm's tumor and cancer metastatic to kidney were excluded.
- Renal Cancer Controls: Renal cancer cases were risk set matched with up to 10 controls for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site. The index date for controls was set as the date at which the follow-up time from cohort entry was the same as the case. The index date was chosen so as to give the control equal follow-up time to that of the case for ascertainment of use of gabapentin.
Period: Overall Study
Arm/Group | Pancreatic Cancer Cases | Pancreatic Cancer Controls | Renal Cancer Cases | Renal Cancer Controls
Started | 3149 | 30026 | 1981 | 19046
Completed | 3149 | 30026 | 1981 | 19046
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pancreatic Cancer Cases: Incident pancreatic cancer, defined as first time pancreatic cancer diagnosis (READ/OXMIS codes) in the GPRD study cohort. Entry into the GPRD study cohort began Jan 1, 1993, or at the time of GPRD registration if after Jan 1, 1993. Subjects were required to have at least 2 years of follow-up prior to the index date. The index date for cases was the date of incident pancreatic cancer diagnosis. Exocrine pancreatic cancer, endocrine pancreatic cancer, and carcinoma in situ were included. Cancer metastatic to the pancreas was excluded.
- Pancreatic Cancer Controls: Pancreatic cancer cases were risk set matched with up to 10 controls for sex, age at cohort entry (within two years), calendar year of cohort entry (within one year), and General Practice site. The index date for controls was set as the date at which the follow-up time from cohort entry was the same as the case. The index date was chosen so as to give the control equal follow-up time to that of the case for ascertainment of use of gabapentin.
- Total: Total of all reporting groups
Arm/Group | Pancreatic Cancer Cases | Pancreatic Cancer Controls | Renal Cancer Cases | Renal Cancer Controls | Total
Number analyzed (Participants) | 3149 | 30026 | 1981 | 19046 | 54202
Age, Customized [Number; unit: Participants] — Number of participants with the indicated age at index date.
  Participants
    <40 years | 18 | 199 | 43 | 446 | 706
    40-49 years | 86 | 897 | 134 | 1348 | 2465
    50-59 years | 367 | 3616 | 355 | 3418 | 7756
    60-69 years | 748 | 7234 | 528 | 5199 | 13709
    70-79 years | 1033 | 10092 | 594 | 5604 | 17323
    >=80 years | 897 | 7988 | 327 | 3031 | 12243
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1603 | 15316 | 759 | 7273 | 24951
  Male | 1546 | 14710 | 1222 | 11773 | 29251
Number of participants with the indicated duration of follow-up from GPRD registration to index date [Number; unit: participants]
  2-3 years | 173 | 1460 | 129 | 1081 | 2843
  4-5 years | 185 | 1509 | 117 | 1135 | 2946
  6-7 years | 237 | 2007 | 141 | 1280 | 3665
  >=8 years | 2554 | 25050 | 1594 | 15550 | 44748
Number of participants with the indicated duration of follow-up from GPRD study cohort entry to ID [Number; unit: participants] — Entry into the GPRD study cohort began Jan 1, 1993, or at the time of GPRD registration if after Jan 1, 1993. Subjects were required to have at least 2 years of follow-up prior to the index date (ID).
  participants
    2-3 years | 446 | 4121 | 286 | 2653 | 7506
    4-5 years | 396 | 3656 | 226 | 2122 | 6400
    6-7 years | 447 | 4213 | 246 | 2338 | 7244
    >=8 years | 1860 | 18036 | 1223 | 11933 | 33052
Number of participants with the indicated body mass index (BMI) [Number; unit: participants] — BMI is calculated as weight in kilograms (between one and three years prior to the index date, closest to 1 year prior to index date) divided by height in meters (one year or longer prior to index date) squared (m^2).
  participants
    <18.5 kg/m^2 | 25 | 203 | 18 | 110 | 356
    18.5 to 24.99 kg/m^2 | 459 | 3678 | 237 | 2236 | 6610
    25 to 29.99 kg/m^2 | 457 | 4250 | 326 | 2938 | 7971
    >=30 kg/m^2 | 291 | 2476 | 250 | 1773 | 4790
    Missing | 1917 | 19419 | 1150 | 11989 | 34475
Number of participants with the indicated smoking status [Number; unit: participants]
  Current Smoker | 731 | 4857 | 476 | 3555 | 9619
  Ex-smoker | 768 | 6626 | 524 | 4589 | 12507
  Never Smoked | 1385 | 15249 | 867 | 9121 | 26622
  Status Unknown | 265 | 3294 | 114 | 1781 | 5454
Number of participants with the indicated medical conditions in Pancreatic Cancer Cases/Controls [Number; unit: participants] — Medical conditions up to the index date by READ/OXMIS codes were analyzed.
  participants
    Diabetes (>=2 years prior to index date [ID]) | 363 | 2137 | 0 | 0 | 2500
    Epilepsy | 53 | 458 | 0 | 0 | 511
    Neuropathic Pain | 737 | 6616 | 0 | 0 | 7353
    Chronic Pancreatitis (>=2 years prior to ID) | 13 | 17 | 0 | 0 | 30
Number of participants with the indicated medical conditions/drug use in Renal Cancer Cases/Controls [Number; unit: participants] — Medical conditions up to the index date by READ/OXMIS codes were analyzed. Drug use up to the index date according to British National Formulary codes was analyzed.
  participants
    Hypertension | 0 | 0 | 1159 | 9113 | 10272
    Diuretic use | 0 | 0 | 875 | 6396 | 7271
    Diabetes | 0 | 0 | 240 | 1598 | 1838
    Epilepsy | 0 | 0 | 33 | 303 | 336
    Neuropathic Pain | 0 | 0 | 428 | 4018 | 4446

OUTCOME MEASURES:

1. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident pancreatic cancer. Gabapentin Exposure Description: Without 2 year lag = Gabapentin prescription from cohort entry to index date. With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer).
Time Frame: The case index date (ID) was the date of incident pancreatic cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control ID was the date at which the follow-up time from his/her cohort entry was the same as that for the case
Population: Cases and controls were drawn from the GPRD study cohort. Entry into the study cohort began Jan 1, 1993, or at the time of GPRD registration if after Jan 1, 1993. Follow-up ended Dec 31, 2008, or earlier if the respective cancer was diagnosed or if the participant left the GPRD for any reason including death.
Measure: Number; unit: participants
Groups:
- Cases: Cases
- Controls: Controls
Arm/Group | Cases | Controls
Number analyzed (Participants) | 3149 | 30026
participants
  Ever (without 2 year lag) | 56 | 253
  Never (without 2 year lag) | 3093 | 29773
  Ever (with 2 year lag) | 24 | 143
  Never (with 2 year lag) | 3125 | 29883
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.04, 95% CI 2-sided [1.51 to 2.75] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0001, Conditional Logistic Regression; Adjusted Odds Ratio = 1.82, 95% CI 2-sided [1.34 to 2.46] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, chronic pancreatitis, neuropathic pain, epilepsy
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0627, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.52, 95% CI 2-sided [0.98 to 2.36] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.2183, Conditional Logistic Regression; Adjusted Odds Ratio = 1.33, 95% CI 2-sided [0.85 to 2.08] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, chronic pancreatitis, neuropathic pain, epilepsy

2. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident pancreatic cancer. Gabapentin Exposure Description: Without 2 year lag = Gabapentin exposure from cohort entry to index date. With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Tertiles without 2 year lag: Tertile 1 (1-2 prescriptions),Tertile 2 (3-8 prescriptions), and Tertile 3 (9-218 prescriptions). Tertile's with 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-10 prescriptions),Tertile 3 (11-191 prescriptions).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 3149 | 30026
participants
  Never (without 2 year lag) | 3093 | 29773
  Tertile 1 (without 2 year lag) | 30 | 99
  Tertile 2 (without 2 year lag) | 12 | 64
  Tertile 3 (without 2 year lag) | 14 | 90
  Never (with 2 year lag) | 3125 | 29883
  Tertile 1 (with 2 year lag) | 14 | 48
  Tertile 2 (with 2 year lag) | 3 | 49
  Tertile 3 (with 2 year lag) | 7 | 46
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.82, 95% CI 2-sided [1.86 to 4.28] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Adjusted Odds Ratio = 2.53, 95% CI 2-sided [1.66 to 3.85] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, chronic pancreatitis, neuropathic pain, epilepsy
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.001, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.75, 95% CI 2-sided [1.51 to 5.03] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0042, Conditional Logistic Regression; Adjusted Odds Ratio = 2.44, 95% CI 2-sided [1.32 to 4.49] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, chronic pancreatitis, neuropathic pain, epilepsy
Statistical Analysis 5: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0645, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.8, 95% CI 2-sided [0.97 to 3.36] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.1232, Conditional Logistic Regression; Adjusted Odds Ratio = 1.65, 95% CI 2-sided [0.87 to 3.11] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, chronic pancreatitis, neuropathic pain, epilepsy
Statistical Analysis 7: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3160, Conditional Logistic Regression; Unadjusted Odds Ratio = 0.55, 95% CI 2-sided [0.17 to 1.78] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.2234, Conditional Logistic Regression; Adjusted Odds Ratio = 0.48, 95% CI 2-sided [0.15 to 1.57] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, chronic pancreatitis, neuropathic pain, epilepsy
Statistical Analysis 9: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3071, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.35, 95% CI 2-sided [0.76 to 2.42] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.6062, Conditional Logistic Regression; Adjusted Odds Ratio = 1.17, 95% CI 2-sided [0.65 to 2.11] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, diabetes, chronic pancreatitis, neuropathic pain, epilepsy
Statistical Analysis 11: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.5205, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.31, 95% CI 2-sided [0.58 to 2.97] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 12: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.8042, Conditional Logistic Regression; Adjusted Odds Ratio = 1.11, 95% CI 2-sided [0.48 to 2.57] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, diabetes, chronic pancreatitis, neuropathic pain, epilepsy

3. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident pancreatic cancer. Gabapentin Exposure Description: Without 2 year lag = Gabapentin exposure from cohort entry to index date. With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Tertile's without 2 year lag: Tertile 1 (0.01 - 1.55 months), Tertile 2 (1.56 - 6.44 months), and Tertile 3 (6.45 - 78.36 months). Tertile's with 2 year lag: Tertile 1 (0.01 - 1.78 months), Tertile 2 (1.79 - 7.20 months), and Tertile 3 (7.21 - 64.13 months).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 3149 | 30026
participants
  Never (without 2 year lag) | 3093 | 29773
  Tertile 1 (without 2 year lag) | 28 | 83
  Tertile 2 (without 2 year lag) | 14 | 79
  Tertile 3 (without 2 year lag) | 14 | 91
  Never (with 2 year lag) | 3125 | 29883
  Tertile 1 (with 2 year lag) | 13 | 44
  Tertile 2 (with 2 year lag) | 4 | 47
  Tertile 3 (with 2 year lag) | 7 | 52
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Unadjusted Odds Ratio = 3.15, 95% CI 2-sided [2.04 to 4.86] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Adjusted Odds Ratio = 2.88, 95% CI 2-sided [1.85 to 4.46] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0015, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.75, 95% CI 2-sided [1.47 to 5.13] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0053, Conditional Logistic Regression; Adjusted Odds Ratio = 2.45, 95% CI 2-sided [1.31 to 4.62] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0777, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.68, 95% CI 2-sided [0.94 to 2.99] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.1762, Conditional Logistic Regression; Adjusted Odds Ratio = 1.5, 95% CI 2-sided [0.83 to 2.69] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 7: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.6990, Conditional Logistic Regression; Unadjusted Odds Ratio = 0.82, 95% CI 2-sided [0.29 to 2.28] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.5274, Conditional Logistic Regression; Adjusted Odds Ratio = 0.72, 95% CI 2-sided [0.26 to 2.01] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 9: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3245, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.34, 95% CI 2-sided [0.75 to 2.39] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.6388, Conditional Logistic Regression; Adjusted Odds Ratio = 1.15, 95% CI 2-sided [0.64 to 2.07] — [estimate comment as in outcome 2, analysis 10]
Statistical Analysis 11: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.796, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.11, 95% CI 2-sided [0.49 to 2.51] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 12: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.8772, Conditional Logistic Regression; Adjusted Odds Ratio = 0.94, 95% CI 2-sided [0.41 to 2.15] — [estimate comment as in outcome 2, analysis 12]

4. Primary Outcome: Number of Pancreatic Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident pancreatic cancer. Gabapentin Exposure Description: Without 2 year lag = Gabapentin exposure from cohort entry to index date. With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Tertile's without 2 year lag: Tertile 1 (0.01 - 33.6 grams), Tertile 2 (33.7 - 185.0 grams), and Tertile 3 (185.1 - 7500.2 grams). Tertile's with 2 year lag: Tertile 1 (0.01 - 39.0 grams), Tertile 2 (39.1 - 210.0 grams), and Tertile 3 (210.1 - 5623.8 grams).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 3149 | 30026
participants
  Never (without 2 year lag) | 3093 | 29773
  Tertile 1 (without 2 year lag) | 28 | 88
  Tertile 2 (without 2 year lag) | 14 | 74
  Tertile 3 (without 2 year lag) | 14 | 91
  Never (with 2 year lag) | 3125 | 29883
  Tertile 1 (with 2 year lag) | 11 | 46
  Tertile 2 (with 2 year lag) | 7 | 47
  Tertile 3 (with 2 year lag) | 6 | 50
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.90, 95% CI 2-sided [1.88 to 4.47] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Adjusted Odds Ratio = 2.65, 95% CI 2-sided [1.71 to 4.11] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0212, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.19, 95% CI 2-sided [1.12 to 4.25] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0522, Conditional Logistic Regression; Adjusted Odds Ratio = 1.95, 95% CI 2-sided [0.99 to 3.81] — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0337, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.87, 95% CI 2-sided [1.05 to 3.32] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0947, Conditional Logistic Regression; Adjusted Odds Ratio = 1.64, 95% CI 2-sided [0.92 to 2.95] — [estimate comment as in outcome 2, analysis 6]
Statistical Analysis 7: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3928, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.42, 95% CI 2-sided [0.64 to 3.16] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.6502, Conditional Logistic Regression; Adjusted Odds Ratio = 1.21, 95% CI 2-sided [0.54 to 2.72] — [estimate comment as in outcome 2, analysis 8]
Statistical Analysis 9: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3275, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.34, 95% CI 2-sided [0.75 to 2.39] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.6365, Conditional Logistic Regression; Adjusted Odds Ratio = 1.15, 95% CI 2-sided [0.64 to 2.08] — [estimate comment as in outcome 2, analysis 10]
Statistical Analysis 11: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.9858, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.01, 95% CI 2-sided [0.42 to 2.41] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 12: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.7671, Conditional Logistic Regression; Adjusted Odds Ratio = 0.87, 95% CI 2-sided [0.36 to 2.12] — [estimate comment as in outcome 2, analysis 12]

5. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Exposure to Gabapentin
Description: Incident renal cancer. Gabapentin Exposure Description: Without 2 year lag = Gabapentin prescription from cohort entry to index date. With 2 year lag = Gabapentin prescription from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer).
Time Frame: The case index date (ID) was the date of incident renal cancer diagnosis ascertained in the GPRD study cohort 1995-2008. The matched control ID was the date at which the follow-up time from his/her cohort entry was the same as that for the case.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 1981 | 19046
participants
  Ever (without 2 year lag) | 32 | 166
  Never (without 2 year lag) | 1949 | 18880
  Ever (with 2 year lag) | 13 | 76
  Never (with 2 year lag) | 1968 | 18970
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0031, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.79, 95% CI 2-sided [1.22 to 2.63] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0095, Conditional Logistic Regression; Adjusted Odds Ratio = 1.68, 95% CI 2-sided [1.13 to 2.49] — Comparison: "Ever (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, hypertension, diuretic use, diabetes, neuropathic pain, and epilepsy
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0970, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.65, 95% CI 2-sided [0.91 to 2.99] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.1123, Conditional Logistic Regression; Adjusted Odds Ratio = 1.63, 95% CI 2-sided [0.89 to 2.97] — Comparison: "Ever (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, hypertension, diuretic use, diabetes, neuropathic pain, and epilepsy

6. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Number of Gabapentin Prescriptions
Description: Incident renal cancer. Gabapentin Exposure Description: Without 2 year lag = Gabapentin exposure from cohort entry to index date. With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Tertiles without 2 year lag: Tertile 1 (1-2 prescriptions),Tertile 2 (3-8 prescriptions), and Tertile 3 (9-218 prescriptions). Tertile's with 2 year lag: Tertile 1 (1-2 prescriptions), Tertile 2 (3-10 prescriptions),Tertile 3 (11-191 prescriptions).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 1981 | 19046
participants
  Never (without 2 year lag) | 1949 | 18880
  Tertile 1 (without 2 year lag) | 16 | 58
  Tertile 2 (without 2 year lag) | 11 | 55
  Tertile 3 (without 2 year lag) | 5 | 53
  Never (with 2 year lag) | 1968 | 18970
  Tertile 1 (with 2 year lag) | 6 | 27
  Tertile 2 (with 2 year lag) | 4 | 28
  Tertile 3 (with 2 year lag) | 3 | 21
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0012, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.53, 95% CI 2-sided [1.44 to 4.44] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0034, Conditional Logistic Regression; Adjusted Odds Ratio = 2.34, 95% CI 2-sided [1.32 to 4.14] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, hypertension, diuretic use, diabetes, neuropathic pain, and epilepsy
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0856, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.18, 95% CI 2-sided [0.9 to 5.32] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, hypertension, diuretic use, diabetes, neuropathic pain, and epilepsy
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0996, Conditional Logistic Regression; Adjusted Odds Ratio = 2.14, 95% CI 2-sided [0.87 to 5.28] — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 5: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0563, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.89, 95% CI 2-sided [0.98 to 3.63] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0896, Conditional Logistic Regression; Adjusted Odds Ratio = 1.77, 95% CI 2-sided [0.92 to 3.43] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, hypertension, diuretic use, diabetes, neuropathic pain, and epilepsy
Statistical Analysis 7: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.5308, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.4, 95% CI 2-sided [0.49 to 4.01] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.5458, Conditional Logistic Regression; Adjusted Odds Ratio = 1.39, 95% CI 2-sided [0.48 to 4.02] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, hypertension, diuretic use, diabetes, neuropathic pain, and epilepsy
Statistical Analysis 9: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.7744, Conditional Logistic Regression; Unadjusted Odds Ratio = 0.87, 95% CI 2-sided [0.35 to 2.19] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.6999, Conditional Logistic Regression; Adjusted Odds Ratio = 0.83, 95% CI 2-sided [0.33 to 2.11] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)". Adjusted for smoking, BMI, hypertension, diuretic use, diabetes, neuropathic pain, and epilepsy
Statistical Analysis 11: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.6528, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.32, 95% CI 2-sided [0.39 to 4.47] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 12: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.6722, Conditional Logistic Regression; Adjusted Odds Ratio = 1.3, 95% CI 2-sided [0.38 to 4.47] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)". Adjusted for smoking, BMI, hypertension, diuretic use, diabetes, neuropathic pain, and epilepsy

7. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Duration of Exposure to Gabapentin
Description: Incident renal cancer. Gabapentin Exposure Description: Without 2 year lag = Gabapentin exposure from cohort entry to index date. With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Tertile's without 2 year lag: Tertile 1 (0.01 - 1.55 months), Tertile 2 (1.56 - 6.44 months), and Tertile 3 (6.45 - 78.36 months). Tertile's with 2 year lag: Tertile 1 (0.01 - 1.78 months), Tertile 2 (1.79 - 7.20 months), and Tertile 3 (7.21 - 64.13 months).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 1981 | 19046
participants
  Never (without 2 year lag) | 1949 | 18880
  Tertile 1 (without 2 year lag) | 15 | 44
  Tertile 2 (without 2 year lag) | 10 | 67
  Tertile 3 (without 2 year lag) | 7 | 55
  Never (with 2 year lag) | 1968 | 18970
  Tertile 1 (with 2 year lag) | 6 | 23
  Tertile 2 (with 2 year lag) | 3 | 31
  Tertile 3 (with 2 year lag) | 4 | 22
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p < 0.0001, Conditional Logistic Regression; Unadjusted Odds Ratio = 3.24, 95% CI 2-sided [1.79 to 5.85] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0005, Conditional Logistic Regression; Adjusted Odds Ratio = 2.9, 95% CI 2-sided [1.59 to 5.28] — [estimate comment as in outcome 6, analysis 2]
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.042, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.54, 95% CI 2-sided [1.03 to 6.25] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0603, Conditional Logistic Regression; Adjusted Odds Ratio = 2.4, 95% CI 2-sided [0.96 to 5.98] — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 5: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3762, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.35, 95% CI 2-sided [0.69 to 2.65] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.4073, Conditional Logistic Regression; Adjusted Odds Ratio = 1.33, 95% CI 2-sided [0.68 to 2.63] — [estimate comment as in outcome 6, analysis 6]
Statistical Analysis 7: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.9294, Conditional Logistic Regression; Unadjusted Odds Ratio = 0.95, 95% CI 2-sided [0.29 to 3.12] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.9875, Wilcoxon (Mann-Whitney); Adjusted Odds Ratio = 0.99, 95% CI 2-sided [0.3 to 3.29] — [estimate comment as in outcome 6, analysis 8]
Statistical Analysis 9: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.66, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.19, 95% CI 2-sided [0.54 to 2.63] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.8110, Conditional Logistic Regression; Adjusted Odds Ratio = 1.1, 95% CI 2-sided [0.5 to 2.45] — [estimate comment as in outcome 6, analysis 10]
Statistical Analysis 11: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3336, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.7, 95% CI 2-sided [0.58 to 4.96] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 12: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.3782, Conditional Logistic Regression; Adjusted Odds Ratio = 1.63, 95% CI 2-sided [0.55 to 4.84] — [estimate comment as in outcome 6, analysis 12]

8. Primary Outcome: Number of Renal Cancer Cases and Matched Controls With the Indicated Cumulative Dose of Gabapentin
Description: Incident renal cancer. Gabapentin Exposure Description: Without 2 year lag = Gabapentin exposure from cohort entry to index date. With 2 year lag = Gabapentin exposure from cohort entry to 2 years prior to index date (to control for prediagnostic prescribing for pain symptoms possibly related to cancer). Tertile's without 2 year lag: Tertile 1 (0.01 - 33.6 grams), Tertile 2 (33.7 - 185.0 grams), and Tertile 3 (185.1 - 7500.2 grams). Tertile's with 2 year lag: Tertile 1 (0.01 - 39.0 grams), Tertile 2 (39.1 - 210.0 grams), and Tertile 3 (210.1 - 5623.8 grams).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 1981 | 19046
participants
  Never (without 2 year lag) | 1949 | 18880
  Tertile 1 (without 2 year lag) | 9 | 45
  Tertile 2 (without 2 year lag) | 17 | 63
  Tertile 3 (without 2 year lag) | 6 | 58
  Never (with 2 year lag) | 1968 | 18970
  Tertile 1 (with 2 year lag) | 5 | 24
  Tertile 2 (with 2 year lag) | 5 | 26
  Tertile 3 (with 2 year lag) | 3 | 26
Statistical Analysis 1: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0841, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.89, 95% CI 2-sided [0.92 to 3.88] — Comparison: "Tertile 1 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 2: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.1313, Conditional Logistic Regression; Adjusted Odds Ratio = 1.75, 95% CI 2-sided [0.85 to 3.63] — [estimate comment as in outcome 6, analysis 2]
Statistical Analysis 3: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.1488, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.03, 95% CI 2-sided [0.78 to 5.34] — Comparison: "Tertile 1 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 4: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.1495, Conditional Logistic Regression; Adjusted Odds Ratio = 2.05, 95% CI 2-sided [0.77 to 5.46] — [estimate comment as in outcome 6, analysis 3]
Statistical Analysis 5: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0013, Conditional Logistic Regression; Unadjusted Odds Ratio = 2.44, 95% CI 2-sided [1.42 to 4.22] — Comparison: "Tertile 2 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 6: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.0026, Conditional Logistic Regression; Adjusted Odds Ratio = 2.34, 95% CI 2-sided [1.35 to 4.07] — [estimate comment as in outcome 6, analysis 6]
Statistical Analysis 7: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.2421, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.78, 95% CI 2-sided [0.68 to 4.69] — Comparison: "Tertile 2 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 8: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.2899, Conditional Logistic Regression; Adjusted Odds Ratio = 1.7, 95% CI 2-sided [0.64 to 4.53] — [estimate comment as in outcome 6, analysis 8]
Statistical Analysis 9: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.9723, Conditional Logistic Regression; Unadjusted Odds Ratio = 0.99, 95% CI 2-sided [0.42 to 2.29] — Comparison: "Tertile 3 (without 2 year lag)" and "Never (without 2 year lag)"
Statistical Analysis 10: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.8206, Conditional Logistic Regression; Adjusted Odds Ratio = 0.91, 95% CI 2-sided [0.39 to 2.13] — [estimate comment as in outcome 6, analysis 10]
Statistical Analysis 11: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.8135, Conditional Logistic Regression; Unadjusted Odds Ratio = 1.15, 95% CI 2-sided [0.35 to 3.82] — Comparison: "Tertile 3 (with 2 year lag)" and "Never (with 2 year lag)"
Statistical Analysis 12: Comparison: Cases vs Controls; Test type: Superiority or Other; p = 0.8173, Conditional Logistic Regression; Adjusted Odds Ratio = 1.15, 95% CI 2-sided [0.34 to 3.86] — [estimate comment as in outcome 6, analysis 12]

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | Pancreatic Cancer Cases | Pancreatic Cancer Controls | Renal Cancer Cases | Renal Cancer Controls
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.